CLINICAL TRIAL: NCT00137761
Title: A Phase II Study of Docetaxel in Combination With ZD 1839 (IRESSA) in Previously Treated Patients With Metastatic Pancreatic Cancer
Brief Title: Docetaxel in Combination With Iressa in Previously Treated Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Matthew Kulke, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-173
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Metastatic Pancreatic Carcinoma
Keywords: Pancreatic Carcinoma; Iressa; Docetaxel
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gefitinib; Docetaxel

INTERVENTIONS:
Drug: ZD 1839 — Taken orally once daily
  Other Names: Iressa
Drug: Docetaxel — Given intravenously once weekly for 2 out of 3 weeks

SUMMARY:
The purpose of this study is to find out what activity the combination of docetaxel and Iressa have against metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Iressa will be taken orally once daily without interruption. Docetaxel will be administered intravenously once weekly for two out of every three weeks. Patients will also receive dexamethasone the night prior, morning of, and the evening after docetaxel treatment to help prevent an allergic reaction.

Every week that chemotherapy is given, blood tests and vital signs will be taken.

After the first 6 weeks of therapy a CT scan (or other radiological procedure) will be done to assess the progress of the disease. If the cancer is responding to the treatment and no unacceptable side effects have occured, treatment with Iressa and docetaxel will continue.

CT scans (or other radiological procedure) will be performed at week 12 and every 9 weeks thereafter to monitor the progress of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic carcinoma (excluding pancreatic endocrine tumors); histologic confirmation of either the primary or metastatic site.
* ECOG performance status of < 1
* > 4 weeks since completion of previous chemotherapy
* > 4 weeks since participation in any investigational drug study
* Peripheral neuropathy of grade < 1
* Patients must have failed a gemcitabine-containing regimen administered in the metastatic, adjuvant, or locally advanced setting.
* Absolute neutrophil count (ANC) > 1,500/mm3
* Hemoglobin > 9.0gm/dl
* Platelets > 100,000/mm3
* Total bilirubin < 2.0mg/dl
* AST and alkaline phosphatase < 5 x upper limit of normal (ULN)
* Albumin > 2.5gm/dl
* CA 19-9 > 1.5 x ULN

Exclusion Criteria:

* Prior therapy with taxane or with epidermal growth factor receptor (EGFR) inhibitors
* More than one prior chemotherapy treatment
* Clinically significant cardiac disease
* Major surgery within 4 weeks of the start of study treatment
* Evidence of central nervous system (CNS) metastases or carcinomatous meningitis or history of uncontrolled seizures, central nervous system disorders.
* Uncontrolled serious medical or psychiatric illness
* Pregnant or breast-feeding women
* Other active malignancy
* Inability to swallow tablets or evidence of a gastrointestinal malabsorption syndrome
* Known severe hypersensitivity to Iressa
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St. John's wort.
* History of severe hypersensitivity reaction to drugs formulated with polysorbate 80
* Any evidence of clinically active interstitial lung disease
* Ascites requiring paracentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-10; Primary Completion 2007-06 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To determine the response rate of Iressa and docetaxel in patients with advanced pancreatic cancer following failure of gemcitabine-based therapy | 3 years

SECONDARY OUTCOMES:
To determine the safety, radiologic response rate, progression-free survival and overall survival of patients treated with Iressa and docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kulke, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts